CLINICAL TRIAL: NCT00854841
Title: Randomized, Open Label Study of Dasatinib (100mg qd) vs. High-Dose Imatinib (600mg) in Patients With Chronic Phase CML Who Have Had Suboptimal Response After 3-18 Months of Therapy With Imatinib (400mg)
Brief Title: The Randomized Study of Dasatinib and High-Dose Imatinib (600mg) in Suboptimal Responder
Status: Available | Type: Expanded Access
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Jooseop Chung/Professor, Pusan National University Hospital
Other Study IDs: CA180-257; KCML02
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; suboptimal response; dasatinib; imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; Imatinib Mesylate

INTERVENTIONS:
Drug: Dasatinib and Imatinib — Dasatinib Dasatinib will be administered orally at a dose of 100 mg QD. During the first month, subjects will be instructed to take dasatinib in the morning.
  Imatinib Imatinib will be administered orally at a dose of 600 mg once daily (QD). Each 600 mg dose should be administered with a meal and taken with a large glass of water. If a scheduled dose is missed for more than 12 hours or dosing is interrupted for toxicity or for any other reason, these doses should be omitted.
  Other Names: Sprycel and Gliveec

SUMMARY:
Research Hypothesis:

Treatment with dasatinib 100 mg QD is superior to imatinib 600 mg QD in terms of complete cytogenetic response (CCyR) in chronic phase (CP) Philadelphia chromosome-positive (Ph+) Chronic Myeloid Leukemia (CML) subjects who are imatinib failures or who have achieved only a suboptimal response after 3-18 months (12-77 weeks) of therapy with imatinib 400 mg.

Primary Objective:

The primary objective of this study is to compare the rate of CCyR of dasatinib (100mg QD) to high-dose imatinib (600 mg QD) therapy at 6 months after randomization in CP Ph+ CML subjects who are imatinib failures or who have achieved only a suboptimal response after 3 - 18 months of imatinib monotherapy at 400 mg/day.

DETAILED DESCRIPTION:
Study Design: Prospective open-label, randomized two arms, multicenter study for the patients with suboptimal response to standard Tx to evaluate efficacy & safety of dasatinib (100mg qd) & imatinib (600mg daily) by CyR & MoR at 3, 6 & 12 months.

* Randomized 1:1
* Crossover to alternate be permitted after confirmed PD at 3M (AP, BC & loss of CHR or MCyR) & absence of any response at 6M.

Duration of Study: Subjects will be treated for up to 12 months, unless disease progression or unacceptable toxicity occurs, the subject withdraws, or the study is discontinued.

Duration of Study: Subjects will be treated for up to 12 months, unless disease progression or unacceptable toxicity occurs, the subject withdraws, or the study is discontinued.

Number of Subjects: A total of 90 subjects will be randomized in 1:1 randomization ratio

Study Population: Subjects 18 years of age or older with CP Ph+ CML and who are imatinib failures or ave achieved only a suboptimal response after 3 - 18 months (12 - 77 weeks) of treatment with 400 mg/day of imatinib monotherapy.

Test Product, Dose and Mode of Administration, Duration of Treatment:

Subjects in the dasatinib arm will begin treatment with dasatinib at an oral dose of 100 mg QD. One dose reduction to 70 mg due to toxicity will be allowed. One dose escalation to 140 mg is allowed under specified circumstances.

Reference Therapy, Dose and Mode of Administration, Duration of Treatment:

Subjects in the imatinib arm will begin treatment with imatinib at an oral dose of 600 mg QD Doses of imatinib can be escalated to 800 mg for patients with inadequate response at 3 months and dose reduction of imatinib is not permitted for any cases of patients.

Criteria for Evaluation:

Efficacy:

* Primary Endpoint: CCyR rate at 6 months after randomization.
* Secondary Endpoints:

  * MMR rates at 3, 6, and 12 months
  * CCyR rates at 3, 6 and 12 months
  * CHR rates at 3, 6and 12 months
  * Time to-, and duration of-, MMR and CCyR
  * Progression free survival (PFS)

Safety:

Adverse experiences associated with dasatinib or imatinib treatment will be reported for all treated subjects. Adverse events will be assessed continuously and graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent, at least 18 years old
2. Adequate hepatic renal function
3. Dasatinib naïve patients
4. Patients with cytogenetically and/or molecularly confirmed Philadelphia chromosome or BCR-ABL positive CP-CML who have been treated with standard dose of imatinib.
5. ECOG status: 0-2
6. And one of following criteria for imatinib suboptimal response 1)CP-CML patients who have failed to achieve a CHR at 3 months or MCyR at 6 months of therapy with imatinib 400mg daily. 2)CP-CML patients who have failed to achieve a CCyR at 12 months with imatinib 400mg daily 3)CP-CML patients who have failed to achieve a MMoR (less than 3 log reduction) at 18 months with imatinib 400mg daily 4)CP-CML patients who have lost molecular response by an increase of BCR-ABL more than 10 times regardless treatment duration.

Exclusion Criteria:

1. Concurrent malignancy
2. Patients who have received SCT
3. Allergy or hypersensitivity reaction to the study drugs
4. Female who are pregnant or breast feeding.
5. T315I mutation
6. History of significant bleeding disorder
7. Women of child bearing potential
8. Uncontrolled or significant CVS disease: IHD. CHF
9. Prior imatinib>400mg, imatinib>18 months
10. Intolerance to imatinib 400mg

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jooseop Chung, MD. PhD, Principal Investigator — Pusan National University Hospital, Korea